CLINICAL TRIAL: NCT06200220
Title: Patients Treated in Real Life With VEnetoclax for WAldenström Macroglobulinemia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: WAVE
Record Dates: First submitted 2023-12-28; First posted 2024-01-10 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2023-12

CONDITIONS: Waldenstrom's Macroglobulinaemia Refractory
MeSH Terms: interventions — venetoclax

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Venetoclax — Observational study

SUMMARY:
Waldenström macroglobulinemia (WM) is an incurable disease. BCL2 antagonist, an important anti-apoptosys molecule, is already approved for the treatment of chronic lymphocytic leukemia (CLL) and acute myeloid leukemia. Recently, a clinical trial including 32 patients with WM treated with Venetoclax showed an overall response rates of 84% and a major response rate of 81%. However, there is no in real life data, in the french population, of the efficiency of Venetoclax in WM. The aim of our multicentric retrospective study is to evaluate the efficiency and tolerance of Venetoclax in WM.

ELIGIBILITY:
Inclusion Criteria:

* Waldenstrom's macroglobulinemia
* Treatment with Venetoclax
* Non opposition

Exclusion Criteria: none

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients from university hospitals in France (16 center)
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2023-12-28 (Actual); Primary Completion 2023-12-28 (Actual); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Efficiency | 2018 to 2025
  ORR, MRR

SECONDARY OUTCOMES:
Tolerance | 2018 to 2025
  Adverse events
Efficiency in specific population | 2018 to 2025
  ORR in CXCR4 mutated patients, ORR in patients previously treated with BTK inhibitors

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Poitiers, Poitiers, France

IPD SHARING:
Plan to Share IPD: No